CLINICAL TRIAL: NCT04912362
Title: Effectiveness of YAG Laser Iridotomy in Preventing Peripheral Anterior Synechia After CO2 Laser-Assisted Sclerectomy Surgery in Primary Open Angle Glaucoma
Brief Title: The Effectiveness of YAG Iridotomy in Preventing Peripheral Anterior Synechia After CLASS in Primary Open Angle Glaucoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2020-527
Record Dates: First submitted 2021-05-31; First posted 2021-06-03 (Actual); Last update posted 2021-06-03 (Actual); Status verified 2020-08

CONDITIONS: Glaucoma, Open-angle
MeSH Terms: conditions — Glaucoma, Open-Angle

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- YAG iridotomy+CLASS (Experimental): YAG iridotomy was performed one week before operation, and then CO2 Laser-Assisted Sclerectomy Surgery was performed
  Interventions: Device: YAG iridotomy
- CLASS (No Intervention): CO2 Laser-Assisted Sclerectomy Surgery only

INTERVENTIONS:
Device: YAG iridotomy — YAG iridotomy was performed one week before operation, and then CO2 Laser-Assisted Sclerectomy Surgery was performed
  Arms: YAG iridotomy+CLASS

SUMMARY:
To investigate the effectiveness of YAG laser iridotomy in preventing peripheral anterior synechia after CO2 Laser-Assisted Sclerectomy Surgery and the long-term effect of reducing intraocular pressure

DETAILED DESCRIPTION:
Group A: YAG laser iridotomy was performed one week before operation, followed by CO2 Laser-Assisted Sclerectomy Surgery; Group B: only CO2 Laser-Assisted Sclerectomy Surgery; The patients were followed up for 1 year to observe and compare the difference of the incidence of peripheral anterior synechia and the effect of long-term intraocular pressure control between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Primary open angle glaucoma patients in Ophthalmic Center;
* Topical use of hypotensive drugs in the treatment of poor or intolerable intraocular pressure control;
* The patients were 18 to 50 years old, regardless of gender;
* Class operation was performed;
* Patients are able and willing to comply with the research guidance and may complete all visits required by the research;
* Informed consent has been signed.

Exclusion Criteria:

* Allergic to any perioperative medication in this study;
* History of ocular trauma;
* Any previous intraocular surgery;
* Gonioscopy showed a narrow angle (Schaffer III or below);
* Secondary glaucoma was diagnosed;
* Optic atrophy caused by other reasons;
* Severe complications such as rupture of posterior capsule and choroidal hemorrhage occurred during operation;
* Patients with severe ocular complications after operation
* The patient's history indicated that he had severe dysfunction of heart, lung, liver and kidney;
* Women in pregnancy, lactation or planned pregnancy;
* The researchers believe that the patient's condition may put the patient at significant risk, may confuse the results of the study, or may significantly interfere with the patient's participation in the study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2023-08 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
Intraocular pressure | 1 year
  Intraocular pressure
Peripheral anterior synechia | 1 year
  Incidence of peripheral anterior synechia

CONTACTS AND LOCATIONS:
Overall Officials: Kaijun Wang, MD, Study Director — 2nd Affiliated Hospital, School of Medicine, Zhejiang University, China
Locations (1):
- Eye center, 2nd Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China